CLINICAL TRIAL: NCT05446246
Title: Predictive Factoris of Failure in Superobese Patients Undergoing Bariatric Surgery
Brief Title: Superobese Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Fabio Medas, Associate Professor, University of Cagliari
Other Study IDs: SuObPat
Record Dates: First submitted 2022-07-01; First posted 2022-07-06 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Superobese patients: Patients with preoperative BMI > 50
  Interventions: Procedure: Bariatric surgery
- Morbidobese patients: Patients with preoperative BMI > 35 and <50
  Interventions: Procedure: Bariatric surgery

INTERVENTIONS:
Procedure: Bariatric surgery — Sleeve gastrectomy

SUMMARY:
Super obesity (SO) is defined as a Body Mass Index (BMI) > 50 kg/m2, and represents the extreme severity of the disease, resulting in an increase in morbidity, mortality, and in poorer quality of life compared with morbid obesity (BMI > 35 and <50 kg/m2).

ELIGIBILITY:
Inclusion Criteria:

* Morbid and superobese patients

Exclusion Criteria:

* Follow up not completed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with BMI > 35
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgical success | 24 months
  BMI <35

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Cagliari, Cagliari, CA, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be made available under reasonable request